CLINICAL TRIAL: NCT03241732
Title: Defining Neurobiological Signatures for Chronic Traumatic Brain Injury Using PET-MRI Technology
Brief Title: PET-MRI in Chronic Traumatic Brain Injury (CTBI)
Acronym: PET-MRIcTBI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 17D.138
Record Dates: First submitted 2017-07-11; First posted 2017-08-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Chronic Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; Brain Trauma; N-acetyl cysteine; Concussion; NAC; Integrative Medicine; Functional magnetic resonance imaging or functional MRI; fMRI; PET; Positron emission tomography; MRI; magnetic resonance imaging; Chronic Traumatic Brain Injury; Neuro Emotive Technique; Subjective Units of Distress (SUDS)
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: There were two intervention arms of the study and a control group. Enrollment for these groups was 120 subjects. One arm focused on adjusting dietary practices to eat foods that have a lower amount of inflammatory molecules that might help reduce overall inflammation in the brain and body. The second arm was the N-acetyl cysteine group to provide patients with a natural supplement that support antioxidants in the body. The third arm of the study is a waitlist control group.
  The fourth arm is a substudy that may re-enroll and re-consent 30 subjects from the original 3 groups, and will recruit additional subjects as needed, who continue to have distress associated with TBI. Subjects will receive sessions with the Neuro Emotive Technique. Participants enrolled in the 4th NET group will be counted in the cohort of 30 for the NET substudy.
Masking Description: This is an Open Label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary (AID) Cohort (Active Comparator): Anti-inflammatory Diet: This arm will focus on adjusting dietary practices to eat foods that have lower amounts of inflammatory foods that might help reduce overall inflammation in the brain and body. This arm will introduce patients to an integrative diet that reduces saturated fats and carbohydrates and emphasizes proteins and omega-3 fats that help reduce inflammation and oxidative damage.
  Interventions: Other: Anti-inflammatory Diet
- Intravenous/Oral NAC Cohort (Active Comparator): N-acetyl Cysteine: This arm provide patients with a natural supplement, n-acetyl cysteine (NAC) which is the N-acetyl derivative of the naturally occurring amino acid, L-cysteine, that supports antioxidants to reduce oxidative damage in the body. NAC is a common over-the-counter supplement.Laboratory studies have suggested that NAC might have a beneficial effect in neurodegenerative disorders such as TBI. Patients in this arm will receive IV NAC once a week plus oral NAC supplement 500 mg twice per day for approximately 3 months until the follow up evaluation.
  Interventions: Dietary Supplement: N-acetyl Cysteine
- Control Cohort (No Intervention): Control Group: Standard of Care Treatment for at least 3 months. After the first 3 month, participants in this arm may crossover to the NAC study arm.
- Neuro Emotive Technique (NET) (Active Comparator): Eligible participants would be evaluated (or re-evaluated) receive neurocognitive tests, and receive baseline PET-MRI and follow up MRI imaging; pre-screening measures distress by the Subjective Units of Distress interview, biofeedback measures of heart rate variability (HRV) and galvanic skin resistance (GSR) and Baseline and post NET blood plasma and serum analysis to measure inflammation and immune function. Participants from the initial study will be re-consented if enrolled in the Neuro Emotive Technique Substudy. SUDS, biofeedback and surveys, MRI imaging and blood draws will be completed again after the 5 NET sessions are complete.
  Interventions: Behavioral: Neuro Emotive Technique

INTERVENTIONS:
Other: Anti-inflammatory Diet — Integrative diet that reduces saturated fats and carbohydrates and emphasizes proteins and omega-3 fats that help reduce inflammation and oxidative damage.
  Arms: Dietary (AID) Cohort
Dietary Supplement: N-acetyl Cysteine — Intravenous and Oral n-acetyl cysteine
  Arms: Intravenous/Oral NAC Cohort
Behavioral: Neuro Emotive Technique — Neuro Emotive Technique sessions
  Arms: Neuro Emotive Technique (NET)

SUMMARY:
Chronic Traumatic Brain Injury (cTBI) symptoms exist in individuals who experienced previous traumatic brain injuries. There are 80-90 thousand individuals who are clinically diagnosed with cTBI, with estimated costs at greater than 60 billion dollars. However, there is a lack of studies using comprehensive diagnostic imaging tools to better understand physiological ramifications of the injury that may help guide therapy. This study uses integrative medicine approaches for persons with cTBI. Another aim of this study will be a continuation of this protocol in an effort to address the ongoing distressing physiological and psychological (anxiety and depression) symptoms associated with cTBI. After completion of the initial 3 study arms, the investigators have amended the protocol to evaluate the physiological and psychological effects and potential symptom improvement of integrative medicine approaches in cTBI patients using the Neuro Emotive Technique (NET). Participants may be re-enrolled in the NET group after completion of participation in the initial study arms. The participants in the NET substudy will be interviewed about Subjective Units of Distress (SUDS) associated with the cTBI event initially and after completion of the NET sessions.

DETAILED DESCRIPTION:
The purpose of this project was to create a comprehensive, extensive, longitudinal diagnostic evaluation of cTBI patients. The evaluation uses a battery of neurocognitive tests, laboratory levels of specific inflammatory compounds, and Positron Emission Tomography (PET) using Fluoro deoxyglucose (FDG) and functional Magnetic Resonance Imaging (fMRI) at baseline and follow up. Participants were evaluated initially with PET, and then at approximately 3 and 6 months to determine the time course of changes within the brain associated with the integrative medicine approach. Three groups of participants were enrolled in the study: a control group, an anti-inflammatory diet group, and an N-acetyl cysteine (NAC) group; NAC is the N-acetyl derivative of the naturally occurring amino acid, L-cysteine. NAC is a common over-the-counter supplement that is also available as an injectable pharmaceutical that protects the liver in cases of acetaminophen overdose. Laboratory studies have displayed some benefits in use of NAC to reduce markers of oxidative damage, protect against cell death, and to increase glutathione in blood, which might be useful in preventing oxidative damage in cTBI patients.

Amendment:

The investigators have amended the original protocol to add a new arm. The purpose of this sub-study is to 30 enroll subjects who have physiological and/or psychological (depression and/or anxiety) symptoms associated with cTBI. Enrollment in this arm of the study would allow for re-enrollment of participants from who still have persistent anxiety, depression symptoms or distress associated with TBI after completing the first phase of this protocol (referenced above). Participants would be evaluated (or re-evaluated) with a battery of neurocognitive tests, including SUDS, NET, and biofeedback measures anxiety levels and receive baseline PET-MRI imaging and follow up functional MRI, neurocognitive tests, including SUDS, NET, and biofeedback measures.

In addition to assessing symptoms associated with TBI, subjects will receive five sessions of Neuro-emotive Technique to address ongoing mood and anxiety symptoms and is conducted by a trained practitioner with clinical credentials in mental health. Subjects who have participated in the initial study will be re-consented if enrolled in the Neuro Emotive Technique Substudy. The investigators will also enroll new subjects with TBI to be enrolled in the NET substudy cohort. In order to gain a greater understanding of the NET program to evaluate whether it reduces anxiety and affects the physiology of the brain in persons with TBI, we believe the potential benefits outweigh the risks. A prescreening interview will be conducted that inquires about current and past treatment for the TBI. In addition, a brief Subjective Units of Distress discussion will assist to determine the extent to which the subject is experiencing distress from TBI or its effects. Upon (re) enrollment and after the completion of the NET sessions. To assess the level of distress, subjects will receive a pre and post biofeedback testing evaluation that measures heart rate variability (HRV) and galvanic skin resistance (GSR) in conjunction with recollection of distress. Pre and post NET blood draw and blood plasma and serum analysis will provide addition information to measure inflammation and immune function for participants in the NET substudy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a history of TBI and complaints of persistent symptoms including cognitive impairment, emotional disturbances, headache, or other symptoms associated with TBI
* Age 18-80 years old
* Patients had no other pre-existing history (i.e. prior to the TBI) of significant medical, neurological, or psychological disorders such as schizophrenia or active substance abuse.
* Minor, stable health problems that should have no substantial effect on cerebral blood flow will be allowed (i.e. controlled hypertension, medication controlled diabetes)
* Able to give informed consent and willing to complete the study
* Patients will be allowed to be taking medications or supplements at the initial intake, but they must be on a stable dose regimen for at least 1 month
* Women of childbearing potential will confirm a negative pregnancy test NET Substudy: Anxiety and/or distress associated with TBI or TBI symptoms by measurement with Subjective Units of Distress, and biofeedback screening

Exclusion Criteria:

* Previous brain surgery.
* Cognitive impairment with significant impact on activities of daily living and/or a score on the Mini-Mental Status examination (or similar) of 25 or lower
* Intracranial abnormalities that may complicate interpretation of the brain scans (e.g., stroke, tumor, vascular abnormality affecting the target area).
* Pregnant or lactating women.
* Enrollment in active clinical trial/ experimental therapy within the prior 30 days.
* Any pre-existing medical conditions that may interfere with cerebral function.
* Subject is unable or unwilling to lie still in the scanner (i.e. due to claustrophobia or weight > 350 pounds)
* Subject has metal in their body or other reason that they cannot undergo magnetic resonance imaging.

Additional exclusionary criteria for the NAC arm:

* Patients taking medications that might interact with the NAC involved in this study will be evaluated on a case by case basis by the PI or study physician.
* Patients that have a history of uncontrolled conditions, e.g.: diabetes, asthma, gastroesophageal reflex disease, or thyroid conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2027-07-08 (Estimated); Study Completion 2027-07-08 (Estimated)

PRIMARY OUTCOMES:
Fluorodeoxyglucose positron emission tomography (FDG-PET). | Baseline in the primary study for waitlist and control groups, not in the NET substudy.
  To measure inflammation and oxidative damage in the brain.
Functional magnetic resonance imaging (fMRI). | NET Substudy: Baseline, 90 ± 30 days and 180 ± 30 days.
  This scan will be used to assess functional connectivity, tractography, and brain volume.

SECONDARY OUTCOMES:
Heart rate variability | Screening at Baseline, and if enrolled 90 ± 30 days and if in waitlist 180 ± 30 days
  NET Substudy: This assessment is a Biofeedback evaluation to measure the physiologic level of distress experienced.
Galvanic Skin Temperature | Screening at Baseline, and if enrolled 90 ± 30 days and if in waitlist 180 ± 30 days
  NET Substudy: This assessment is a Biofeedback evaluation to measure the physiologic level of distress experienced.
Subjective Units of Distress | Screening at Baseline, and if enrolled 90 ± 30 days and if in waitlist 180 ± 30 days
  NET Substudy: This assessment is a Likert scale that identifies the level of psychological distress experienced.
Blood plasma and serum analysis | Screening at Baseline, and if enrolled 90 ± 30 days
  NET Substudy: Blood draw to evaluate cytokine profile analysis to measure inflammation.
Blood plasma and serum analysis | Follow up, post NET enrolled 90 ± 30 days
  NET Substudy: Blood draw to evaluate T Cell profile analysis will measure immune function.
Rivermead Post-Concussion Symptoms Questionnaire. | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire will be used as one of the quality of life measures for the study.
Beck Depression Inventory (BDI). | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire will be used as one of the psychological evaluation questionnaires for the study.
Speilberger State Trait Anxiety Inventory (STAI). | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire will be used as one of the psychological evaluation questionnaires for the study.
Profile of Moods Scale (POMS). | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire will be used as one of the psychological evaluation questionnaires for the study.
Epworth Sleepiness Scale. | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire will be used as one of the quality of life measures for the study.
Mayo-Portland Adaptability Inventory-4. | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire will be used as one of the quality of life measures for the study.
Delis Kaplan Executive Function System (DKEFS) color-word interference. | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire may be used as one of the cognitive testings for the study.
Trails A & B. | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire may be used as one of the cognitive testings for the study.
Forward and reverse digit span. | Baseline, 90 ± 30 days and 180 ± 30 days.
  This assessment questionnaire may be used as one of the cognitive testings for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B. Newberg, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Villanova, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Muller JJ, Wang R, Milddleton D, Alizadeh M, Kang KC, Hryczyk R, Zabrecky G, Hriso C, Navarreto E, Wintering N, Bazzan AJ, Wu C, Monti DA, Jiao X, Wu Q, Newberg AB, Mohamed FB. Machine learning-based classification of chronic traumatic brain injury using hybrid diffusion imaging. Front Neurosci. 2023 Aug 24;17:1182509. doi: 10.3389/fnins.2023.1182509. eCollection 2023. PMID 37694125
- [Derived] Vedaei F, Mashhadi N, Zabrecky G, Monti D, Navarreto E, Hriso C, Wintering N, Newberg AB, Mohamed FB. Identification of chronic mild traumatic brain injury using resting state functional MRI and machine learning techniques. Front Neurosci. 2023 Jan 9;16:1099560. doi: 10.3389/fnins.2022.1099560. eCollection 2022. PMID 36699521
- [Derived] Teichner EM, You JC, Hriso C, Wintering NA, Zabrecky GP, Alavi A, Bazzan AJ, Monti DA, Newberg AB. Alterations in cerebral glucose metabolism as measured by 18F-fluorodeoxyglucose-PET in patients with persistent postconcussion syndrome. Nucl Med Commun. 2021 Jul 1;42(7):772-781. doi: 10.1097/MNM.0000000000001397. PMID 33660691

DOCUMENTS (1):
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT03241732/ICF_003.pdf